CLINICAL TRIAL: NCT03127618
Title: Lorlatinib - PF-06463922
Status: Approved for marketing | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B746
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Lorlatinib

SUMMARY:
Lorlatinib expanded access program

ELIGIBILITY:
Inclusion Criteria:

* Adult, Senior

Exclusion Criteria:

-

Min Age: 18 Years
Age Groups: Adult, Older Adult